CLINICAL TRIAL: NCT01062438
Title: Genomic Study of Metastatic Osteosarcoma Using Next-Generation Sequencing Technology
Brief Title: Studying DNA in Tumor Tissue Samples From Patients With Localized or Metastatic Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST10B3; COG-AOST10B3 (Other: Children's Oncology Group); CDR0000665327 (Other: Clinical Trials.gov); NCI-2011-02210 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Sarcoma
Keywords: localized osteosarcoma; metastatic osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Gene Expression Profiling; Gene Rearrangement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: mutation analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at DNA in tumor tissue samples from patients with localized or metastatic osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the genomic expression profile in tumor tissue samples from patients with localized or metastatic osteosarcoma using transcriptome sequencing.
* Identify activating and loss of function mutations and gene rearrangement in these tumor tissue samples using transcriptome sequencing.
* Identify candidate genes that are important in osteosarcoma and tumorigenesis using genome partition strategies for genomic DNA sequencing.
* Identify which mutations are associated with outcome.
* Establish which mutations are also found in germ line DNA that predispose the patient to osteosarcoma.

OUTLINE: DNA and RNA from banked tumor tissue samples and DNA from paired blood samples are analyzed in sequencing studies using next-generation sequencing technology. The sequencing data from these tumor samples are matched to the Human RefSeq (for transcriptome sequencing) and normal human genome in the public databases and to the patient's germ line sequence to identify constitutional and somatic mutations.

Clinical information that is associated with each sample (i.e., age, tumor site, size, primary metastases, response to chemotherapy, surgical remission, follow-up time, and treatment protocol) is also collected, if available.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized or metastatic osteosarcoma
* Banked snap-frozen tumor tissue samples and paired blood DNA samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of localized or metastatic osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Genomic expression profile in osteosarcoma tumor samples using transcriptome sequencing
Identification of activating and loss of function mutations and gene rearrangement using transcriptome sequencing
Mutations associated with outcome
Mutations also found in germ line DNA that predispose the patient to osteosarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Javed Khan, MD, Principal Investigator — NCI - Oncogenomics Section